CLINICAL TRIAL: NCT01898169
Title: Evaluation of Plasma Nicotine, Carbon Monoxide, Heart Rate, Craving and Withdrawal After Acute Use of the NJOY King E-Cigarette in the Clinic, Following a One-Week Actual Use Pilot Study
Brief Title: Evaluation of Short-term Safety and Use Patterns of an Electronic Nicotine Delivery System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LA Clinical Trials (Other)
Collaborators: NJOY, Inc. (Industry)
Responsible Party: Principal Investigator, Mitchell Nides, Ph.D., President, LA Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NJ-001 LACT; ISRCTN95345566 (Other: ISRCTN)
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NJOY King 26 mg nicotine Electronic Nicotine Delivery System (Experimental)
  Interventions: Other: NJOY King 26 mg nicotine Electronic Nicotine Delivery System

INTERVENTIONS:
Other: NJOY King 26 mg nicotine Electronic Nicotine Delivery System — NJOY® King ENDS, menthol or nonmenthol, ad libitum use for 1 week NJOY® King ENDS, menthol or nonmenthol, 2 series of puffs, with a 30-second interpuff interval in each series and 1 hour between the first puff in each series.

SUMMARY:
Electronic Nicotine Delivery Systems (ENDS), commonly referred to as electronic cigarettes have gained in popularity over the last several years. The technology used to manufacture ENDS has been evolving rapidly with a variety of delivery mechanisms, nicotine content, e-liquids and flavorings. Only in the last few years have researchers begun to examine the health risks and benefits, nicotine blood levels, patterns of use, likability, and craving and withdrawal relief of ENDS. These studies have shown great variability in nicotine delivery, effects on heart rate, and relief of craving or withdrawal among various ENDS brands among tobacco cigarette smokers.

This study will test a new generation ENDS, the NJOY King Bold (NJOY, Scottsdale, AZ). It is a single use unit that resembles a traditional cigarette and delivers approximately 150 puffs. The cartridge inside contains 26 milligrams of nicotine.

Our primary objective is to evaluate the short-term effects of using the NJOY Kings ENDS on heart rate, carbon monoxide and blood nicotine levels and well as on craving for cigarettes and nicotine withdrawal. Our secondary objective is to evaluate the subject's usage patterns for cigarettes and NJOY King ENDS during a one-week period in which they can use each freely.

The study includes three visits to the clinic spaced approximately one week apart. Subjects who pass the screening visit will return to the clinic for Visit 2 in which they will sample the NJOY King ENDS for about 20 minutes before taking home enough to last till Visit 3, one week later. They will be instructed to use as many or as few as they like during the week. Subjects will keep a daily diary of number of tobacco cigarettes smoked and number of e-cigarette puffs taken. Subjects will return to the clinic for Visit 3 after 12 hours of abstinence from any form of nicotine in order to assure that they have no nicotine left in their bloodstream. Eligible subjects will then participate in two series of 10 puffs of NJOY Kings spaced one hour apart. During the 2.5 hours of the testing day, the following will be measured: 1) heart rate, 2) carbon monoxide, 3)blood will be sampled for nicotine levels, 4) craving for cigarettes and nicotine withdrawal symptoms will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy cigarette smokers
2. Not trying or planning to quit
3. >10 factory-produced cigarettes/day for previous year
4. Breath carbon monoxide level of >10 ppm at screening

Exclusion Criteria:

1. Pregnancy or lactation
2. Abuse of drugs other than tobacco
3. Use of any prescription psychoactive medications within 14 days
4. Use of ENDS within 14 days
5. Use of any nicotine replacement within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Change in blood nicotine levels | Change from baseline at Visit 3 to 5, 10, 15 and 30 minutes after each of two series, spaced one hour, apart of 10 puff from the NJOY King at Visit 3
  Note: Visit 3 can occur up to 28 days after the Screening Visit
Change in average cigarettes smoked per day | The baseline week compared to the week testing the NJOY Kings in the "real world"
  Subjects will have a one weeks supply of NJOY Kings to use as they like. Mean cigarettes per day during the "actual use week" will be compared to the mean cigarettes per day for the baseline week (which is one week before the "actual use" week)
Average NJOY Kings puffs used per day | Day 1 through Day 6 of the of testing the NJOY Kings in the "real world"
  Mean number of puffs per day of NJOY King ENDS used during Day 1 through Day 6 of the actual use week which can begin 1 to 3 weeks after the Screening Visit

CONTACTS AND LOCATIONS:
Overall Officials: MITCHELL NIDES, Ph.D., Principal Investigator — LA Clinical Trials
Locations (1):
- LA Clinical Trials, Burbank, California, United States